CLINICAL TRIAL: NCT03946709
Title: Mirror Neurons in Older Participants (Project MNOP): Acute Effects of Action Observation on Muscle Strength/Weakness and Neurophysiological Factors in Older Adults
Brief Title: Mirror Neurons in Older Participants
Acronym: MNOP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 risk in older adults.
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Matt Stock, Assistant Professor, University of Central Florida
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SBE-18-14657
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Muscle Weakness; Dynapenia; Sarcopenia
MeSH Terms: conditions — Muscle Weakness; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Muscle strength condition (Other)
  Interventions: Other: Action Observation
- Muscle weakness condition (Other)
  Interventions: Other: Action Observation
- Control (No Intervention)

INTERVENTIONS:
Other: Action Observation — Strength, voluntary activation, and cortical responses to three conditions will be measured: 1) action observation of very strong, forceful contractions of the hand and wrist flexors 2) action observation of very weak, feeble contractions of the hand and wrist flexors 3) no action observation. Experimental conditions will be randomized and counterbalanced.
  Arms: Muscle strength condition; Muscle weakness condition

SUMMARY:
A critical problem facing aging adults is muscle weakness. Whereas scientists have traditionally attributed the loss of muscle strength with aging to muscle atrophy, emerging evidence suggests that impairments in the neuromuscular system's ability to voluntarily generate force plays a more central role than previously appreciated. One area that has not yet been investigated includes the role that observing another's actions - thereby activating mirror neurons - plays in muscle force generation. Therefore, the purpose of this study is to examine the acute effects of action observation on muscular strength, voluntary muscle activation, and cortical excitability and inhibition in older adults.

DETAILED DESCRIPTION:
A critical problem facing aging adults is muscle weakness. Whereas scientists have traditionally attributed the loss of muscle strength with aging to atrophic effects, emerging evidence suggests that impairments in the neuromuscular system's ability to voluntarily generate force plays a more central role than previously appreciated. One area that has not yet been investigated includes the role that observing another's actions - thereby activating mirror neurons - plays in muscle force generation. Therefore, the purpose of this study is to examine the acute effects of action observation on muscular strength, voluntary activation, and cortical excitability and inhibition in older adults. Following a thorough familiarization visit, twenty-five men and women ≥60 years of age will complete three action observation sessions in a randomized, counterbalanced manner: 1) observation of very strong hand/wrist contractions, 2) observation of very weak hand/wrist contractions, and 3) a control condition. Maximal voluntary contractions (MVCs) of the wrist flexors will be performed before and after observation sessions. Percent voluntary activation will be determined via the interpolated twitch technique. Single-pulse transcranial magnetic stimulation (TMS) and electromyographic (EMG) recordings from the flexor carpi radialis and first dorsal interosseous will be used to quantify cortical excitability and inhibition, via motor evoked potential amplitude and silent period duration, respectively. The hypothesis of this study is that observation of strong muscle contractions will acutely increase muscle strength, and such changes will be facilitated by enhanced corticospinal excitability and decreased inhibition. In contrast, it is hypothesized that observation of very weak contractions will cause no such efforts or even acute muscle weakness. Collectively, we propose that manipulation of mirror neurons is a worthwhile strategy for clinicians hoping to induce neuromuscular adaptations in older adults, particularly in settings where movement of a joint is painful or infeasible (e.g., bedrest or immobilization).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women ≥60 years of age

Exclusion Criteria:

* Neuromuscular disease (e.g. Parkinson's, MS, ALS)
* Metabolic disease (e.g. diabetes, thyroid disorder, metabolic syndrome)
* Arthritis in the upper limbs (hands, arms, shoulders)
* Trouble using or controlling one's muscles
* History of cancer
* History of stroke
* History of heart attack
* Use of an assistive walking device or other mobility aids
* Physician mandated contraindication to exercise within the last 6 months
* Epilepsy or history of convulsions/seizures
* History of fainting or syncope
* History of head trauma that was diagnosed as concussion or was associated with loss of consciousness
* History of hearing problems or tinnitus
* Cochlear implants
* Implanted metal in the brain, skull, or elsewhere in the body
* Implanted neurotransmitter
* Cardiac pacemaker or intracardiac lines
* Medication infusion device
* Past problems with brain stimulation
* Past problems with MRI
* Use of muscle relaxants or benzodiazepines
* Allergy to rubbing alcohol
* Any other health related illnesses that would prohibit a participant from physical performance testing
* Lack of transportation to and from the laboratory

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | 5 minutes
  Isometric muscle strength of the non-dominant hand and wrist flexors will be assessed during maximal voluntary contractions (MVCs).

SECONDARY OUTCOMES:
Voluntary Activation | 5 minutes
  Percent voluntary activation will be quantified during the MVCs to determine each participant's ability to maximally activate their wrist flexor muscles voluntarily.
Corticospinal excitability | 5 minutes
  Transcranial magnetic stimulation will be used to quantify corticospinal excitability throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Matt S. Stock, Ph.D., Principal Investigator — University of Central Florida
Locations (1):
- UCF Neuromuscular Plasticity Laboratory, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harmon KK, Girts RM, Pagan JI, Rodriguez G, Stock MS. The acute effects of action observation on muscle strength/weakness and corticospinal excitability in older adults. Exp Brain Res. 2022 Jun;240(6):1801-1810. doi: 10.1007/s00221-022-06370-2. Epub 2022 Apr 29. PMID 35488129